CLINICAL TRIAL: NCT02654925
Title: Myeloid to Adipocyte Transdifferentiation in Human Cells
Acronym: MYTH
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-1779; UL1TR001082 (NIH)
Record Dates: First submitted 2016-01-07; First posted 2016-01-13 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Young Men: men 21-40 years of age
  Interventions: Procedure: Adipose Tissue Biopsy
- Young Women: women 21-40 years of age; young women will be premenopausal and eumenorrheic, not on hormonal contraceptive therapy.
  Interventions: Procedure: Adipose Tissue Biopsy
- Older Men: men 55-100 years of age
  Interventions: Procedure: Adipose Tissue Biopsy
- Older Women: women 55-100 years of age; older women will be postmenopausal who are at least 12 months past the final menstrual period (FMP).
  Interventions: Procedure: Adipose Tissue Biopsy

INTERVENTIONS:
Procedure: Adipose Tissue Biopsy

SUMMARY:
In order to design new programs to help prevent weight gain, promote successful and sustainable weight loss, and help treat diseases related to obesity, the investigators need a better understanding of why accumulating fat in certain regions of the body is bad for health. It is known that not all fat cells are the same, but it was recently discovered that some fat cells may arise from stem cells that come from the bone marrow (bone marrow progenitors), a previously unrecognized origin. This discovery has been paradigm shifting, because dogma has long held that all white fat cells arise from fat tissue resident mesenchymal stem cells. This is also important because fat cells arising from the bone marrow lineage may be linked to worse health outcomes. The aim of this study is to determine if cells that were not previously believed to contribute to fat generation in humans are indeed capable of becoming fat cells. To answer this question the investigators will take samples of cells from the blood and the fat tissue of younger and older men and women, isolate the cells that came from the bone marrow and grow them in culture to determine if they will turn into fat cells. The results of this investigation may reveal potential mechanistic targets for future therapies to reduce the negative health outcomes associated with obesity related chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 21-40 y or 55-100 y;
* Older women will be postmenopausal who are at least 12 months past the final menstrual period (FMP);
* Young women will be premenopausal and eumenorrheic, not on hormonal contraceptive therapy;
* Body Mass Index (BMI) 22-35 kg/m2;
* Non-active to moderately active (vigorous exercise ≤ 3 days/wk lasting < 30 min).

Exclusion Criteria:

* Immunosuppression therapy;
* On blood thinners, aspirin, or NSAIDs that cannot be withheld for the biopsy;
* Prior history of allergies to local anesthetics;
* Current use of hormones, or glucose lowering medication;
* Currently engaged in a vigorous exercise or diet program;
* Currently gaining or losing weight or using weight loss drugs;
* Type 2 diabetes (past/current diagnosis or treatment);
* Diagnosis of uncontrolled metabolic disorders (e.g., thyroid);
* History of severe obesity BMI ≥ 40 or significant weight loss (≥ 50 lbs);
* Postmenopausal - hormonal menopausal therapy use currently or in the previous 6 months;
* Premenopausal - irregular menstrual cycles defined as 2 or more missed cycles in the previous year, pregnant or planning to become pregnant during the study timeline (urine pregnancy test will be performed before DEXA [dual energy x-ray absorptiometry] scan is completed).

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2016-03; Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Adipogenic potential as measured by Oil Red-O staining (quantification by absorbance). | Within 60 days of biopsy
Adipocyte specific gene expression will be measured by qPCR (quantitative polymerase chain reaction) to confirm adipocyte status. | Sample collection within 60 days of biopsy, batched analysis completed depending on enrollment.

SECONDARY OUTCOMES:
Assessment of the fraction of myeloid cells that become 'mesenchymal-like' (CD45-/CD14-/CD34+) (CD: cluster of differentiation) after fibrin culture by flow cytometry. | Within 2 weeks of biopsy
Progenitor cell proliferation capacity as measured by BrdU (bromodeoxyuridine) incorporation | Within 60 days of biopsy
In vivo adipogenesis in the Matrigel plug will be assessed by immunohistochemistry (IHC) for adipocyte (e.g., adiponectin) and nuclear markers (e.g., DAPI). | Samples will be collected within 60 days of biopsy, batched sample analysis will occur dependent on subject enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Gavin, PhD, Principal Investigator — University of Colorado Denver Anschutz Medical Campus
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No